CLINICAL TRIAL: NCT05924711
Title: "Association Between the Treatment of Peri-implantitis and the Resolution of Maxillary Sinusitis: a Case-control Study".
Brief Title: "Association of Peri-implantitis and Maxillary Sinusitis: a Case-control Study".
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Ramón Pons Calabuig, Principal investigator, Clinical Professor, Universitat Internacional de Catalunya
Other Study IDs: PER-ECL-2023-02
Record Dates: First submitted 2023-06-06; First posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Peri-Implantitis; Sinusitis; Sinusitis, Acute; Sinusitis, Chronic; Implant Infection; Dental Implant Failure Nos
MeSH Terms: conditions — Peri-Implantitis; Sinusitis; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: The case group will consist of 20 patients who will have implants diagnosed with peri-implantitis, according to the 2017 World Workshop Classification case definition.
  Interventions: Other: Retrospective analysis of demographic and radiographic data previously obtained from the patient.
- Control group: The control group will include 20 subjects who will have implants with peri-implant health according to the 2017 World Workshop Classification case definition.
  Interventions: Other: Retrospective analysis of demographic and radiographic data previously obtained from the patient.

INTERVENTIONS:
Other: Retrospective analysis of demographic and radiographic data previously obtained from the patient. — The patient's demographic data obtained previously by anamnesis and clinical examination will be retrospectively analyzsed. On the other hand, a radiographic evaluation including analysis of the implants, adjacent teeth and maxillary sinuses/sinus membranes shall be performed using computer software.

SUMMARY:
Scientific evidence regarding the influence of peri-implantitis on Schneider's membrane thickening is scarce and limited. Similarly, to date, there is no literature documenting the resolution of implant-associated maxillary sinusitis with peri-implantitis after treatment of peri-implantitis or removal of the implant. Therefore, the aim of this case-control study is to investigate the association between peri-implantitis and maxillary sinusitis. On the other hand, the changes that occur at the level of the maxillary sinus membrane after treatment of peri-implantitis or after implant explantation will be evaluated.

DETAILED DESCRIPTION:
Background Scientific evidence regarding the influence of peri-implantitis on Schneider's membrane thickening is scarce and limited. Similarly, to date, there is no literature documenting the resolution of implant-associated maxillary sinusitis with peri-implantitis after treatment of peri-implantitis or removal of the implant.

Objectives Therefore, the aim of this case-control study is to investigate the association between peri-implantitis and maxillary sinusitis. On the other hand, the changes that occur at the level of the maxillary sinus membrane after treatment of peri-implantitis or after implant explantation will be evaluated.

Hypothesis H01: The presence of implants placed in the posterior maxillary region affected by peri-implantits is associated with sinus membrane thickening or maxillary sinusitis.

H11: The presence of implants placed in the posterior maxillary region affected by peri-implantits is not associated with sinus membrane thickening or maxillary sinusitis.

H02: Treatment of peri-implantitis in implants placed in the posterior maxillary region can resolve maxillary sinusitis or reduce sinus membrane thickening.

H12: Treatment of peri-implantitis on implants placed in the posterior maxillary region cannot resolve maxillary sinusitis or reduce sinus membrane thickening.

Material and methods Study design The study will present a case-control design. Patients will be retrospectively recruited from a private clinic exclusively dedicated to periodontics and implantology (Clínica CICOM, Badajoz, Spain).

Study setting The study will be conducted in a private practice associated with the Universitat Internacional de Catalunya (UIC). The study protocol and informed consent will be reviewed by the Ethics Committee of the Universitat Internacional de Catalunya (UIC, Barcelona, Spain) and the Declaration of Helsinki, 1975, revised in 2013, will be followed.

Study population All patients included in the study will sign the corresponding informed consent forms for each of the treatments received, as well as for the use of their demographic and radiographic data for scientific purposes.

The subjects recruited will be edentulous (partial/total) patients who previously had implants placed in the posterior region of the maxilla for oral rehabilitation. The case group will consist of 20 patients who will have implants diagnosed with peri-implantitis while in the control group the 20 subjects included will have implants with peri-implant health.

Demographic data

A set of demographic data shall be obtained and recorded:

1. Sex (M/F)
2. Age (years)
3. History of periodontal disease (according to the latest classification of periodontal disease from the report of the "Consensus report of workgroup 4 of the 2017 World Workshop on the Classiﬁcation of Periodontal and Peri-Implant Diseases and Conditions): severity (I, II, III and IV), grade (A, B and C) and extent (localized, generalized or inicisive-molar pattern).
4. Type of edentulism: partial or total.
5. Number of implants per patient
6. Smoking (heavy smoker >10 cig/day, light smoker <10 cig/day, ex-smoker 0 cig/day, or non-smoker 0 cig/day).
7. Position of the implants: premolar region or molar region of the maxilla.
8. Time in function (years)
9. Implant diagnosis (according to the latest classification of periodontal disease from the "Consensus report of workgroup 4 of the 2017 World Workshop on the Classiﬁcation of Periodontal and Peri-Implant Diseases and Conditions): peri-implant health, mucositis or peri-implantitis.
10. Previous history of maxillary sinusitis
11. Implant-related variables:

    1. Implant placed with horizontal bone augmentation (Y/N) or with sinus lift (Y/N and lateral/transcrestal window).
    2. Implant system (diameter, length and type of connection)
    3. Implant macro-design (transmucosal or bone level)

       Radiographic analysis Images of the included patients will be obtained with the CBCT-ICAT Model 17-19 (Imaging Sciences International LLC, Hatfield, PA, USA). The parameters were set as 16x13 mm in width and depth, 120 kVp, 20.27 mAs, scan time 14.7 seconds, resolution at 0.25 voxels and field of view varying according to the region scanned. Radiographic evaluation will include analysis of implants, adjacent teeth and maxillary sinuses/sinus membranes.

       Radiographic analysis of the implants

       A pre-calibrated examiner (RP) will analyze each of the implants included in the study using the coDiagnostiX software (Implant planning Software, Dental Wings GmbH, Chemnitz, Germany). The following parameters will be evaluated:

       - Peri-implant radiographic bone loss: assessed at 4 sites per implant (mesial, distal, vestibular and palatal). The distance from the implant platform to the first bone-to-implant contact (Bone-to-implant contact) in mm shall be measured.

       These radiographic measurements shall be repeated again in the case group subjects after the peri-implantitis has been treated. The time between treatment and the re-evaluation tac shall be at least 6 months.

       Radiographic evaluation of adjacent teeth A pre-calibrated examiner (RP) will analyze each adjacent tooth for the presence of periapical lesions or carious lesions using the coDiagnostiX software (Implant planning Software, Dental Wings GmbH, Chemnitz, Germany). This is recorded as presence or absence.

       Radiographic evaluation of the maxillary sinus

       A pre-calibrated examiner (BA) will analyze each maxillary sinus using Dolphin 3D Images software. The following parameters will be evaluated:
       * Distance from the apex of the implant to the maxillary sinus: measured from the apical portion of the maxillary cortex to the apex of the implant following the longitudinal axis of the implant, measured in mm.
       * Sinus membrane thickening (sagittal direction): measured from the cortical bone of the raised sinus floor to the upper margin of the sinus mucosa at the point of greatest thickening, measured in mm.
       * Thickening of the sinus membrane (coronal): measured from the cortical bone of the floor of the raised sinus to the upper margin of the sinus mucosa at the point of greatest thickening, measured in mm.
       * Volume of the maxillary sinus occupied by the sinus membrane: the total volume of the sinus membrane (cm3 and %) shall be calculated compared to the total volume of the maxillary sinus.

       These radiographic measurements will be repeated again in the case group subjects after treatment of peri-implantitis or after explantation of implants in more advanced cases. The time between treatment and the re-evaluation tac will be at least 6 months.

       In addition, the following information shall be obtained for each maxillary sinus and sinus membrane:
       * Mucosal inflammation: 0 (clear sinus), 1 (mild membrane thickening) and 2 (moderate membrane thickening).
       * Sinus ostium patency: 0 (patent ostium) or 1 (obstructed ostium).
       * Implant-to-sinus ratio: 0 (distance between implant apex and sinus with presence of cancellous bone and cortical bone between implant and sinus), 1 (implant contacts the sinus cortical bone) and 2 (implant is partially inserted into the sinus).

       Case definition of peri-implantitis Peri-implantitis will be defined according to the 2017 Word Workshop of Periodontal and Peri-implant diseases. Therefore, the case definition applied will be as follows: presence of bleeding and/or oozing on soft probing (∼0.2N), peri-implant probing depths of ≥6 mm, bone levels ≥3 mm apical to the most coronal portion of the intra-osseous part of the implant according to periapical radiography.

       Morphology and severity of peri-implant bone defect The characterization of peri-implant defects will be based on the morphology of the defect (Classes I-III) and severity (grades L-M-A), as previously proposed. Briefly, according to morphology it will be classified as follows Class I: infra-bony defect (Class IA: buccal dehiscence, Class IB: 2- to 3-wall defect), Class II: supra-crestal/horizontal defect, and Class III: combined defect (Class IIIA: buccal dehiscence + horizontal bone loss, Class IIIB: 2- to 3-wall defect + horizontal bone loss, Class IIIC: circumferential defect + horizontal bone loss). In terms of severity, implants shall be classified as follows: Mild (L): 3 to 4 mm/ <25% of implant length, Moderate (M): 4 to 5 mm/≥25% to 50% of implant length, and Advanced(A): >6 mm/ >50% of implant length.

       Statistical analysis The statistical package (SPSS 15.0, SPSS Inc., Chicago, IL, USA, STATISTICS, version 7.1StatSoft, Inc., USA AND R 2.14.0) will be used to analyze the data. Pearson's correlation test will be applied for the assessment of confounding factors.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 18-80 years of age
* Patients with implants in the posterior sector of the upper jaw
* Dental implant carriers with a follow-up of more than 5 years
* Patients who have undergone a CT scan for the evaluation of these implants or for other reasons

Exclusion Criteria:

* Patients with uncontrolled systemic disease
* Pregnant or lactating patients
* Heavy smokers (HS)
* Patients with uncontrolled or active periodontal disease in need of periodontal treatment
* Patients with zygomatic or pterygoid implants
* Patients taking medications known to modify bone metabolism or who have degenerative bone disease (hyperparathyroidism, osteoporosis), vitamin D, patients who have taken antibiotics, NSAIDs or corticosteroids for more than two weeks in the last 3 months prior to the examination.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes — Men and women between 18-80 years of age
Study Population: All patients included in the study signed the corresponding informed consent forms for each of the treatments received, as well as for the use of their demographic and radiographic data for scientific purposes.
  The subjects recruited will be edentulous (partial/total) patients who previously had implants placed in the posterior region of the maxilla for oral rehabilitation. The case group will consist of 20 patients who will have implants diagnosed with peri-implantitis while in the control group the 20 subjects included will have implants with peri-implant health.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2023-07-05 (Estimated); Study Completion 2023-07-15 (Estimated)

PRIMARY OUTCOMES:
Sinus membrane thickening changes after peri-implantitis treatment | 6 months
  Sagital and coronal linear measurements of membrane thickening

SECONDARY OUTCOMES:
Severity of peri-implantitis in implants with maxillary sinusitis | 1 month
  Linear measurements at 4 implant sites measured on the available CT scans of the patients
Volume dimensional changes of the sinus membrane | 1 month
  Total membrane occupancy inside the sinus and amount of sinus free of occupation

CONTACTS AND LOCATIONS:
Overall Officials: Jose Nart, PhD, Study Chair — UIC
Locations (2):
- Spain (2):
  - Universitat Internacional de Catalunya (UIC), Sant Cugat del Vallès, Barcelona
  - Ramon Pons, Barcelona

IPD SHARING:
Plan to Share IPD: No
Data collected from patients may only be processed by the research team of this study and will not be shared with other researchers.